CLINICAL TRIAL: NCT02973373
Title: MRI of the Chest Under High Frequency Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Beigelman-Aubry Catherine, MD, University of Lausanne Hospitals
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-HFV
Record Dates: First submitted 2016-11-17; First posted 2016-11-25 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Non-invasive Ventilation; High-frequency Ventilation; Healthy Volunteer
Keywords: MRI; Chest; Apnea
MeSH Terms: conditions — Apnea | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI with HF-NIV (Experimental): Intervention: Acquisition of MRI with High-Frequency non-invasive ventilation (HF-NIV)
  Interventions: Device: MRI with High-frequency non-invasive ventilation
- MRI without HF-NIV (Active Comparator): Intervention: MRI without High-Frequency non-invasive ventilation (HF-NIV)
  Interventions: Other: MRI without High-frequency non-invasive ventilation

INTERVENTIONS:
Device: MRI with High-frequency non-invasive ventilation — MRI performed under high-frequency non-invasive ventilation
  Arms: MRI with HF-NIV
Other: MRI without High-frequency non-invasive ventilation — MRI performed without High-frequency non-invasive ventilation
  Arms: MRI without HF-NIV

SUMMARY:
The purpose of the study is to evaluate the benefit on image quality of MRI of the chest performed under high frequency non-invasive ventilation. This technique indeed allows to generate an apnea duration of several minutes with acquisitions performed at full inspiration. This study will be applied on healthy subjects.

DETAILED DESCRIPTION:
High frequency ventilation (HF-V) has been applied by using a non-invasive interface allowing to obtain a prolonged apnea in awaken subjects. Such an application should be of interest for MRI taking into account its susceptibility to motion of the chest and the imperfect techniques of respiratory gating that are usually performed at end expiration. The purpose of this study is to assess the benefit on image quality of different sequences performed with and without the device in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjets : normal respiratory function and no known lung disease
* Age >=18y

Exclusion Criteria:

• Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Image quality assessment (soapbubble, maximum of first derivative, signal to noise, contrast to noise) | within 2 weeks after MRI acquisition
  Image quality and artefacts will be evaluated and compared without and with the device. Sharpness of the interfaces between vessels and lung will be evaluated with the Soapbubble software (Etienne et al., Magn Reson Med. 2002 Oct;48(4):658-66). The interface between diaphragm and lung will be evaluated with the maximum of the first derivative (Tibiletti et al., Magn Reson Med. 2016 Mar;75(3):1324-32). Signal to noise and contrast to noise will be measured within regions of interest in the image.

SECONDARY OUTCOMES:
Heart and coronary arteries evaluation (soapbubble, signal to noise, contrast to noise) | within 2 weeks after MRI acquisition
  The potential benefit on the exploration of the heart and coronary arteries will be assessed. Sharpness of the coronary arteries with respect to the neighbouring tissue will be evaluated with the Soapbubble software (Etienne et al., Magn Reson Med. 2002 Oct;48(4):658-66). Signal to noise and contrast to noise will be measured within regions of interest in the image.
Synchronization of the acquisition | during the MRI examination
  The possibility of synchronizing the MRI acquisition with the ventilation system will be explored with the aim to eliminate residual diaphragmatic motion and evaluate the potential additional benefit in terms of image quality and artefacts will be evaluated.
Subjective tolerance (questionnaire) | at the end of the MRI examination
  Subjective tolerance of MRI examination under HF-NIV (questionnaire). Participants will fill the questionnaire right after the examination end.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine I Beigelman-Aubry, MD, Principal Investigator — University Hospitals Lausanne Switzerland
Locations (1):
- University Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delacoste J, Dournes G, Dunet V, Ogna A, Noirez L, Simons J, Long O, Berchier G, Stuber M, Lovis A, Beigelman-Aubry C. Ultrashort echo time imaging of the lungs under high-frequency noninvasive ventilation: A new approach to lung imaging. J Magn Reson Imaging. 2019 Dec;50(6):1789-1797. doi: 10.1002/jmri.26808. Epub 2019 May 28. PMID 31136048